CLINICAL TRIAL: NCT04751448
Title: COLON MD: Colon Cancer Longitudinal Study of the Microbial Metabolites and Dietary Factors That Influence Response to Treatment
Brief Title: COLON-MD: Colon Cancer Longitudinal Study
Acronym: COLON-MD
Status: Recruiting | Type: Observational
Sponsor: Baylor Research Institute (Other)
Collaborators: Baylor University (Other)
Responsible Party: Sponsor
Other Study IDs: 017-342
Record Dates: First submitted 2021-02-02; First posted 2021-02-12 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Colon Cancer
Keywords: FOLFOX Treatment
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool sample kit, Tissue at time of surgery, blood draw(2 vials) at specific times up to 5 times.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational: All patients going on study will be put in the observational grouping for blood and tissue collection with option for stool collection.

SUMMARY:
The goal of this proposal is to identify how the composition of the gut microbiome and diet interact to impact chemotherapy-induced diarrhea incidence and severity.

DETAILED DESCRIPTION:
In this longitudinal observational study patients will supply samples of their gut microbiome prior to scheduled colonoscopy or surgery along with dietary intake and blood samples; the relative abundance of microbes from those samples along with dietary data will be used to predict the presence or absence and severity of chemotherapy-induced diarrhea. Microbiome and diet based predictions from blinded samples will be combined to map the diet-microbiome changes during treatment to the changes in immune markers and risk of chemotherapy-induced diarrhea.

ELIGIBILITY:
Inclusion Criteria:

* Colon cancer diagnosis
* Age >18 and < or equal to 79.
* Ability to perform informed consent
* FOLFOX treatment expected

Exclusion Criteria:

* Not Pregnant
* Does not have Lynch syndrome or FAP diagnosis.
* Inability to perform inform consent
* inability to comply with follow up program
* history of prior colon cancer diagnosis
* previous treatment with antibiotics in the last month.
* previous bowel resection.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Colon cancer patient, prior to surgery or prior to treatment start
Sampling Method: Probability Sample
Enrollment: 11 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Microbiome-Based Prediction of Chemotherapy-induced Diarrhea in Colon Cancer | 3 years
  Microbiome analysis from at least 112 blinded samples will be conducted from fecal samples to determine sensitivity, specificity and accuracy (reported as percentage) of a microbiome-based predictor of chemotherapy-induced diarrhea in colon cancer.

SECONDARY OUTCOMES:
Dietary-Based Prediction of Chemotherapy-induced Diarrhea in Colon Cancer | 3 years
  Dietary analysis from at least 112 blinded surveys will be conducted using food frequency questionnaires (DHQ-III) plus 24 hour recalls collected during treatment to determine sensitivity, specificity and accuracy (reported as percentage) of a dietary-based predictor of chemotherapy-induced diarrhea in colon cancer.

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor Research Institute, Temple, Texas, United States

DOCUMENTS (1):
  • Study Protocol (2020-10-21): https://cdn.clinicaltrials.gov/large-docs/48/NCT04751448/Prot_000.pdf